CLINICAL TRIAL: NCT00089154
Title: A Phase II Study of Thrice Weekly Apolizumab in Patients With Chronic Lymphocytic Leukemia : CRC Master Protocol
Brief Title: Apolizumab in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01454; OSU 0410; CLLRC-OSU-0410; CDR0000378072; OSU-0410; NCI-6257; R21CA091564 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Noncontiguous Stage II Small Lymphocytic Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage III Small Lymphocytic Lymphoma; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — apolizumab

ARMS (1):
- Treatment (apolizumab) (Experimental): Patients receive apolizumab IV over 2-4 hours on days 1, 2, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: apolizumab; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: apolizumab — Given IV
  Other Names: 1D1O Anti-lymphoma Antibody; MOAB 1D10; MoAb Hu1D10; Monoclonal antibody 1D10; Monoclonal Antibody Hu1D10
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying how well apolizumab works in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma. Monoclonal antibodies such as apolizumab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate and progression-free survival rate in patients with relapsed or refractory chronic lymphocytic leukemia (CLL) or noncontiguous stage II or stage III or IV small lymphocytic lymphoma treated with apolizumab.

II. Determine the safety of this drug, in terms of the frequency and severity of treatment-related adverse events, in these patients.

SECONDARY OBJECTIVES:

I. Determine clinical response to apolizumab varies by genetic subtype of CLL. II. Determine if pharmacokinetic clearance is truly predicted by 1D10 antigen density on the individual patient CLL cell and how apolizumab clearance correlates with response and selected toxicities observed.

III. To determine the importance of reactive oxygen species and specific signaling pathways in promoting apolizumab-mediated apoptosis in vitro and in vivo in primary CLL cells and if this correlates with clinical response to therapy.

IV. To determine the cellular properties which convey resistance to apolizumab in CLL in vivo.

OUTLINE: This is a multicenter study.

Patients receive apolizumab IV over 2-4 hours on days 1, 2, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 week, at 1 and 2 months, every 3 months for 1 year, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed hematologic malignancy of 1 of the following histologies:

  * Chronic lymphocytic leukemia (CLL)
  * Small lymphocytic lymphoma (SLL)

    * Noncontiguous stage II or stage III or IV disease
* Received >= 1 form of prior immunotherapy or chemotherapy

  * Completed therapy at least 4 weeks ago
* Requires therapy (unless early bone marrow transplantation is planned), as indicated by 1 of the following criteria:

  * Progressively worsening disease (symptoms increasing in severity by 1 toxicity criterion over a period of >= 2 weeks)
  * Progressively worsening anemia or thrombocytopenia
  * Progressively worsening lymphadenopathy
  * Massive splenomegaly or hypersplenism
  * Hyperlymphocytosis (WBC > 200,000/mm^3) OR lymphocyte doubling time < 12 months
  * Marrow failure due to marrow infiltration by leukemia or lymphoma
* Leukemia cells must express 1D10 antigen > 2 times mean fluorescent intensity of the control by flow cytometry of blood or bone marrow cells
* Performance status - ECOG 0-2
* At least 2 years
* Platelet count >= 50,000/mm^3 (transfusion independent)
* Bilirubin =< 3 mg/dL (unless due to tumor involvement)
* Creatinine =< 2.0 mg/dL
* No decompensated congestive heart failure
* No unstable angina
* No myocardial infarction within the past 6 months not corrected by surgery or percutaneous transluminal coronary angioplasty
* No active infection requiring oral or IV antibiotics
* No other malignancy that limits life expectancy to < 2 years or that requires active anticancer therapy within 4 weeks of study entry
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study treatment
* Recovered from prior immunotherapy
* More than 3 months since prior alemtuzumab or rituximab
* No prior apolizumab
* Recovered from prior chemotherapy
* More than 4 weeks since prior anticancer hormonal therapy
* More than 4 weeks since prior anticancer radiotherapy
* More than 4 weeks since prior anticancer surgery
* At least 4 weeks since other prior therapy for CLL or SLL and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-08; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Response rate (CR+PR) | Up to 3 years
Progression-free survival rate | Up to 3 years
Frequency and severity of treatment-related adverse events | Up to 30 days

SECONDARY OUTCOMES:
Pharmacokinetic clearance | Days 1, 2, 3, 5, 8, 15, 22, 26, 27, 29 and 1, 2, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Byrd, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Chronic Lymphocytic Leukemia Research Consortium (CRC), La Jolla, California
  - Ohio State University Medical Center, Columbus, Ohio